CLINICAL TRIAL: NCT05214196
Title: The Effectiveness of Oral Antiseptics on the Intraoral Viral Load of SARS-CoV-2
Brief Title: The Efficacy of Oral Antiseptics Against COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sema Nur Sevinc, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MIC1
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19; Viral load; Antiseptic; Povidone-iodine; Hypochlorous acid
MeSH Terms: conditions — COVID-19 | interventions — Hypochlorous Acid; Povidone-Iodine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hypochlorous acid group (Experimental): The effect of 0.02% Hypochlorous acid solution on viral load was investigated by using 25 COVID-19 patients as an oral antiseptic for 30 seconds.
  Interventions: Drug: Hypochlorous Acid 0.02% Soln,Top (Crystaline) (HClO)
- Povidone-iodine group (Active Comparator): The effect on viral load was investigated by using 0.5% Povidone-iodine solution as an oral antiseptic for 30 seconds in 25 COVID-19 patients.
  Interventions: Drug: Hypochlorous Acid 0.02% Soln,Top (Crystaline) (HClO)
- Saline group (Placebo Comparator): The effect on viral load was investigated by using 0.9% isotonic saline solution as a placebo for 30 seconds in 25 COVID-19 patients.
  Interventions: Drug: Hypochlorous Acid 0.02% Soln,Top (Crystaline) (HClO)

INTERVENTIONS:
Drug: Hypochlorous Acid 0.02% Soln,Top (Crystaline) (HClO) — SARS-CoV-2 sample was obtained from COVID-19 patients by rinsing the mouth and throat with 5 ml of isotonic saline before and 30 minutes after rinsing. In the hypochlorous acid group, 20 ml of HClO was asked to be rinsed in the mouth and throat for 30 seconds in 25 participants. In the povidone-iodine group, 20 ml of PVP-I was asked to be rinsed in the mouth and throat for 30 seconds in 25 participants. In the saline group, 20 ml of saline was asked to be rinsed in the mouth and throat for 30 seconds in 25 participants.
  Other Names: Povidone-iodine 0.5% (Betadine) (PVP-I); Isotonic saline 0.9% (Gifrer)

SUMMARY:
In a study conducted on 75 COVID-19 patients, the effect of SARS-CoV-2 on viral load was investigated as a result of the use of hypochlorous acid and povidone-iodine as an oral antiseptic.

DETAILED DESCRIPTION:
Before and 30 minutes after rinsing with mouth antiseptics, the participants were asked to rinse the mouth and throat for 30 seconds with 0.9% isotonic saline. The sample was sputtered into a sterile plastic container. The participants were grouped according to the type of oral antiseptics used. The effectiveness of SARS-CoV-2 viral load was investigated by rinsing the mouth and throat for 30 seconds with 20 ml of hypochlorous acid, povidone-iodine, and isotonic saline. Viral load was analyzed by RT-PCR analysis. The results were evaluated by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 RT-PCR result,
* Adult hospitalized patient,
* The participants have the physical and psychological ability to follow the instructions in the study.

Exclusion Criteria:

* Patients intubated and supported by a mechanical respirator,
* Severe acute or chronic medical or psychiatric condition,
* History of significant adverse effects following use of oral hygiene products such as toothpaste and mouth rinses,
* Active uncontrolled thyroid disease,
* Developmental/cognitive disability,
* Pregnancy,
* Undergoing radioactive iodine therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
RT-PCR analysis | two weeks
  For the quantitative analysis of the amount of SARS-CoV-2 RNA in the obtained samples, the Real-time Reverse Transcyptase Polymerase Chain Reaction method was used.

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Dilsiz, Prof., Principal Investigator — Atatürk University, Faculty of Dentistry
Locations (1):
- Atatürk University Faculty of Dentistry, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sevinc Gul SN, Dilsiz A, Saglik I, Aydin NN. Effect of oral antiseptics on the viral load of SARS-CoV-2: A randomized controlled trial. Dent Med Probl. 2022 Jul-Sep;59(3):357-363. doi: 10.17219/dmp/150831. PMID 35904769